CLINICAL TRIAL: NCT00921362
Title: Seroquel (Quetiapine Fumarate) InPractice Evaluation Programme
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-NRO-SER-2006/2; SER-01-S-06
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Schizophrenia patients under Seroquel treatment

SUMMARY:
Patients eligible for entry into the study have a diagnosis of schizophrenia defined by Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria and of a chronic or sub-chronic nature.The primary purpose of the study is to observe symptoms changes over 6 months in schizophrenia in patients treated with Seroquel; additionally disease severity and treatment compliance are followed

ELIGIBILITY:
Inclusion Criteria:

* To assess at baseline and after treatment administration the severity of the illness in patients with schizophrenia, using the scores obtained after the application of the CGI scale
* To assess the changes in symptoms of patients treated with Seroquel for 24 weeks, using BPRS (Brief Psychiatry Rating Scale) as measuring tool

Exclusion Criteria:

* All the patients who have a known hypersensitivity to Seroquel /quetiapine or any of its excipients will not be included in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients eligible for entry into the study will have a diagnosis of schizophrenia defined by Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria and of a chronic or sub-chronic nature
Sampling Method: Probability Sample
Enrollment: 1387 (Actual)
Dates: Start 2006-05; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale - BPRS | Monthly at every clinic visit- 7 times

SECONDARY OUTCOMES:
Clinical Global Impression Severity of Illness | Monthly/ at every clinic visit-7 times
CGI-S Clinical Global Impression Improvement CGI -I | Monthly/ at every clinic visit except first visit- 6 times

CONTACTS AND LOCATIONS:
Overall Officials: stina Pentiuc, Med Director, Study Director — AstraZeneca Romania